CLINICAL TRIAL: NCT04280224
Title: Clinical Investigation of Natural Killer Cells Treatment in Pneumonia Patients Infected With 2019 Novel Coronavirus
Brief Title: NK Cells Treatment for COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henan Medical University (Other)
Collaborators: First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK-COVID19
Record Dates: First submitted 2020-02-13; First posted 2020-02-21 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Novel Coronavirus Pneumonia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NK Cells Treatment Group (Experimental): Conventional treatment plus NK cells. Participants will receive conventional treatment plus twice a week of NK cells (0.1-2*10E7 NK cells/kg body weight).
  Interventions: Biological: NK Cells
- Conventional Control Group (No Intervention): Participants will only receive conventional treatment.

INTERVENTIONS:
Biological: NK Cells — twice a week of NK cells (0.1-2*10E7 cells/kg body weight)
  Arms: NK Cells Treatment Group

SUMMARY:
Since december 2019, acute respiratory disease due to 2019 novel coronavirus (2019-nCoV) emerged in Wuhan city and rapidly spread throughout China. There is no confirmed antivirus therapy for 2019-nCoV infection. Natural killer (NK) cells are innate lymphocytes that may serve as useful effectors against danger infection. The purpose of this clinical investigation is to evaluate the safety and efficiency of NK Cells in combination with standard therapy for pneumonia patients infected with 2019-nCoV.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female, aged at 18 years-65 years old
* 2. Pneumonia that is judged by chest radiograph or computed tomography
* 3. Laboratory confirmation of NCP infection by reverse-transcription polymerase chain reaction(RT-PCR) from any diagnostic sampling source

Exclusion Criteria:

* 1. Pregnancy or breastfeeding
* 2. Known HIV, HBV or HCV infection
* 3. Patients with malignant tumor, other serious systemic diseases and psychosis
* 4. Patients who are participating in other clinical trials
* 5. Inability to provide informed consent or to comply with test requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement of clinical symptoms including duration of fever | Measured from day 0 through day 28
  Evaluation of pneumonia improvement
Improvement of clinical symptoms including respiratory frequency | Measured from day 0 through day 28
  Evaluation of pneumonia improvement
Number of participants with treatment-related adverse events evaluated with CTCAE,version 4.0 | Measured from day 0 through day 28
  Safety evaluation

SECONDARY OUTCOMES:
Time of virus nucleic acid test negative | Measured from day 0 through day 28
  Marker for 2019-nCoV
CD4+ and CD8+ T cell count | Measured from day 0 through day 28
  Marker of immunological function
Rate of mortality within 28-days | Day 28
  Marker for efficacy of treatment
Size of lesion area by thoracic imaging | Measured from day 0 through day 28
  Recovery of lung injury

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan, China

IPD SHARING:
Plan to Share IPD: No